CLINICAL TRIAL: NCT01848821
Title: Pilot Study of the Effect of OASIS Ultra on Critical Sized Wound Healing
Brief Title: The Effect of OASIS Ultra on Critical Sized Wound Healing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel Dante Yeh, Trauma & Critical Care Surgeon, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-P-001903/1
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Wound; Infective Wound; Iatrogenic Critical Sized Wound Defects; Wound Healing
Keywords: OASIS ultra; faster healing time; better healing quality; standard of care

STUDY DESIGN:
Intervention Model Description: OASIS
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OASIS half of wound (Other): OASIS will be applied to one half of the wound and standard of care consisting of wound vac only will be applied to the other half.
  Interventions: Device: OASIS Ultra
- Standard therapy half of wound (Other): Standard therapy to half of wound will consistent of non-stick mesh and wound VAC application.
  Interventions: Device: Wound VAC Standard Therapy

INTERVENTIONS:
Device: OASIS Ultra — Porcine derived intestinal submucosa
  Arms: OASIS half of wound
Device: Wound VAC Standard Therapy — Negative pressure wound device aka wound VAC will be placed on the standard therapy half of the wound
  Other Names: Negative Pressure Wound Device
  Arms: Standard therapy half of wound

SUMMARY:
The aim of this study is to evaluate the speed and quality with which OASIS® Ultra (Healthpoint Biotherapeutics; Fort Worth, Texas) increases wound healing in the critical sized defect. The investigators intend on confirming the histological composition of the dermal substitute in order to delineate the amount of cellular recruitment, collagen deposition and neovascularization present compared with control wounds. The investigators hypothesize that OASIS® Ultra will provide a faster healing time as well as the re-establishment of a dermis for further skin graft application. The investigators anticipate that our study will define parameters for the application of OASIS® Ultra as well as potentially demonstrating the advantages in healing time, healed wound quality and hospital stay.

DETAILED DESCRIPTION:
The eligible participants for this study include all patients >18 years with traumatic, infective or iatrogenic critical sized wound defects (50 sq cm or greater) with a quantitative wound culture < 105. Accrual of patients will take place at the Massachusetts General Hospital Churchill Surgical Service. All eligible patients will be identified by physician care givers on the Churchill service. Non-study affiliated physicians will then approach the patient and/or his or her healthcare proxy with a consent form and a direct description of the study. If the patient and/or his or her healthcare proxy agree to proceed with inclusion then the described protocol will be followed.

Patients with the following medical diagnoses will be excluded from the study:

* Wounds that cannot have a negative pressure wound device applied due to anatomical difficulty (i.e. proximity to perineum/anus) or exposed arteries/veins.
* Patients who are DNR/DNI
* Patients who are hemodynamically unstable or requiring pressors
* Patients that are immunodeficient or immunocompromised (ie HIV)
* Patients that have any allergy to porcine products
* Patients that have a religious or ethical necessity to avoid porcine products
* Patients whose wounds are derived from extension of mitotic lesions (ie ulcerative squamous cell carcinoma)
* Patients whose wounds are expected to heal in less than seven days or be ready for skin grafting in less than seven days with standard therapy
* Patients with full thickness burns
* Patients with wound surface area of <50 sq cm
* Pregnant patients (as confirmed by serum or urinary beta-Human Chorionic Gonadotrophin sampling or by History).

Subject Enrollment:

The study will take place between January 1, 2013 (or IRB approval date) and June 30, 2015. The eligible participants for this study include all patients >18 years with traumatic, infective or iatrogenic critical sized wound defects (50 sq cm or greater) with a quantitative wound culture < 105. Accrual of patients will take place at the Massachusetts General Hospital Churchill Surgical Service. All eligible patients will be identified by physician care givers on the Churchill service. Non-study affiliated physicians will then approach the patient and/or his or her healthcare proxy with a descriptive consent form and a verbal explanation of the study. If the patient and/or his or her healthcare proxy agree to proceed with inclusion then the described protocol will be followed.

Consent The consent form is written in non-medical 'lay' terms in order that all non-medical readers may understand the terminologies and ideas. If the patient is non-English speaking then a certified hospital translator will be obtained in order that the written and verbal discussions can be done in the patient's native language for full comprehension. The PHRC policy on Obtaining and Documenting Informed Consent of Subjects who do not Speak English will be followed. For this study, potential subjects will be given a written translation in a language understandable to them of the "short form" or of the entire English version of the consent form approved by the Partners Human Research Committee (PHRC). Once a patient has been identified as eligible for enrollment by a physician on the team, a verbal discussion will be had with the patient using the sections of the consent form ensuring to cover purpose of research, design of research, procedures, risks, benefits, discomforts, benefits, costs, alternatives and number of patients to be enrolled. After identification of eligible patients, verbal explanation of the study parameters while leaving the patient with the consent form to read, 24 hours will be allowed to pass in order that the patient may think about potential questions and/or issues he or she may have with the study. Upon return by a physician not affiliated with the study, they will answer any patient questions or concerns. If the patient is willing to proceed with consent the co-Investigator or principal investigator will be contacted in order that the patient and the investigator may co-sign the consent form. We will ensure that there are contact details on the patient's consent form should they have any questions or issues. If the patient wishes to withdraw consent prior to the completion of the study they will be allowed to do so and the IRB will be contacted for guidance. The informed consent authorizes the use of medical chart information, historical lab values and consent for photography.

The PHRC recommendations regarding categories of surrogates (listed in general order of preference) that may provide consent in writing on behalf of potential subjects incapable of providing informed consent will be followed:

i) court appointed guardian with specific authority to consent to participation in research or authority to make health care decisions for a class of diagnostic and therapeutic decisions inclusive of the proposed research;

ii) health care proxy/person with durable power of attorney with specific authority for making health care decisions inclusive of the proposed research; or

iii) spouse, adult child, or other close family member who knows the subject well and has been involved in their care. Assent of subjects will be a requirement for participation in the research unless the subject is incapable of giving assent due to his/her medical condition. If the individual objects to participation, s/he should not be enrolled. When surrogate consent is relied upon, the Investigator will ensure that the surrogate understands that his or her decisions should be based on "substituted judgment." This means that the decision reflects a potential subject's own views when s/he had the capacity to express them.

The Investigators will document the relationship of the surrogate to the subject in the research record.

ELIGIBILITY:
Inclusion Criteria:

* all patients >18 years
* traumatic, infective or iatrogenic critical sized wound defects (50 sq cm or greater)
* quantitative wound culture < 105.

Exclusion Criteria:

* Wounds that cannot have a negative pressure wound device applied due to anatomical difficulty (i.e. proximity to perineum/anus) or exposed arteries/veins.
* Patients who are DNR/DNI
* Patients who are hemodynamically unstable or requiring pressors
* Patients that are immunodeficient or immunocompromised (ie HIV)
* Patients that have any allergy to porcine products
* Patients that have a religious or ethical necessity to avoid porcine products
* Patients whose wounds are derived from extension of mitotic lesions (ie ulcerative squamous cell carcinoma)
* Patients whose wounds are expected to heal in less than seven days or be ready for skin grafting in less than seven days with standard therapy
* Patients with full thickness burns
* Patients with wound surface area of <50 sq cm
* Pregnant patients (as confirmed by serum or urinary beta-Human Chorionic Gonadotrophin sampling or by History).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dante Yeh, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: wound halves
Groups:
- OASIS: OASIS Ultra (Porcine derived intestinal submucosa) to half of the wound.
  Negative Pressure Wound Therapy (NPWT) aka wound VAC will be placed on the OASIS half of the wound.
- Standard Therapy: Standard therapy to half of wound will consistent of non-adherent dressing and overlying VAC application.
  Negative Pressure Wound Therapy (NPWT) aka wound VAC will be placed on the standard therapy half of the wound.
Period: Overall Study
Arm/Group | OASIS | Standard Therapy
Started | 7; 10 wound halves | 7; 10 wound halves
Completed | 7; 10 wound halves | 7; 10 wound halves
Not Completed | 0; 0 wound halves | 0; 0 wound halves

BASELINE CHARACTERISTICS:
Population: A total of 7 patients with 10 wounds were enrolled in the study.
Units Other Than Participants: Wound halves
Groups:
- Total: Total of all reporting groups
Arm/Group | OASIS Half of Wound | Standard Therapy Half of Wound | Total
Number analyzed (Participants) | 7 | 7 | 7
Number analyzed (Wound halves) | 10 | 10 | 20
Age, Customized [Mean (Standard Deviation); unit: years]
  Years | 51.4 (24.1) | 51.4 (24.1) | 51.4 (24.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 1 | 1 | 1
  Male | 6 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Days from first debridement to OASIS application [Median (Inter-Quartile Range); unit: days] | 6 [4.25 to 6] | 6 [4.25 to 6] | 6 [4.25 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Size From Baseline to Final Wound Evaluation up to 60 Days Later
Description: High-resolution digital photographs of the wound are taken (with a measurement scale included in the picture) at baseline and during serial wound evaluations in the operating room, at the bedside, and in the clinic. The picture is then uploaded into a wound tracing software program (Analyzing Digital images, www.umassk12.net/adki/) and wound area is calculated. Only the Baseline Measure and Final Wound Evaluation are used to calculate the Primary Outcome.
Time Frame: Baseline, Final Wound Evaluation up to 60 Days Later
Measure: Median (Inter-Quartile Range); unit: cm^2
Units Other Than Participants: wound halves
Arm/Group | OASIS | Standard Therapy
Number analyzed (Participants) | 7 | 7
Number analyzed (wound halves) | 10 | 10
cm^2 | -20.7 [-30.3 to -13.8] | -13.9 [-26.3 to -11.]

2. Secondary Outcome: Change in Histological Acute Inflammation Score From Baseline to Skin Grafting Procedure
Description: At baseline and at every dressing change up to the skin grafting procedure, tissue biopsies for histopathological evaluation are obtained using a disposable dermal biopsy punch (8-mm diameter) or scalpel and locations of the biopsy sites within the wound are systematically rotated.
  Only biopsies from the Baseline and Final Skin Grafting Procedure are used to calculate this outcome measure.
  Parameters of acute inflammation (polymorphonuclear neutrophil infiltrate, edema, hemorrhage, and necrosis) were semiquantitatively assessed using a scoring system as follows: 0, non/minimal; 1, mild; 2, moderate, 3, marked. Each parameter was assigned a score, for a minimum and maximum total possible score of 0 and 12. A higher score represents a higher degree of acute inflammation.
Time Frame: Baseline, Final Skin Grafting Procedure
Measure: Median (Inter-Quartile Range); unit: Histolotical Acute Inflammation Score
Units Other Than Participants: wound halves
Arm/Group | OASIS | Standard Therapy
Number analyzed (Participants) | 7 | 7
Number analyzed (wound halves) | 10 | 10
Histolotical Acute Inflammation Score | -2.5 [-3.3 to -1] | 0 [-1.3 to 1.3]

3. Secondary Outcome: Change in Histological Repair Score From Baseline to Skin Grafting Procedure
Description: At baseline and at every dressing change up to the skin grafting procedure, tissue biopsies for histopathological evaluation are obtained using a disposable dermal biopsy punch (8-mm diameter) or scalpel and locations of the biopsy sites within the wound are systematically rotated.
  Parameters of tissue repair (fibroblast proliferation, collagen density, and neovascularization) were semiquantitatively assessed using a scoring system as follows: 0, none/minima; 1, mild; 2, moderate; 3, marked. Each parameter was assigned a score for a total minimum and maximum possible score of 0 and 9. A higher score represents more advanced wound healing.
Time Frame: Baseline, final Skin Grafting procedure
Measure: Median (Inter-Quartile Range); unit: Histological Repair Score
Units Other Than Participants: wound halves
Arm/Group | OASIS | Standard Therapy
Number analyzed (Participants) | 7 | 7
Number analyzed (wound halves) | 10 | 10
Histological Repair Score | 4.5 [-0.25 to 6] | 2.5 [1 to 4.25]

ADVERSE EVENTS:
Arm/Group | OASIS | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
This study is limited by its small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No